CLINICAL TRIAL: NCT05311085
Title: Cytisine and E-cigarettes With Supportive Text-messaging for Smoking Cessation
Brief Title: Cytisine and E-cigarettes With Supportive Text-messaging for Smoking Cessation (Cess@Tion)
Acronym: Cess@Tion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor in Population Health, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/323
Record Dates: First submitted 2021-11-05; First posted 2022-04-05 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; e-cigarette; cytisine; vaping; pragmatic; effectiveness
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — cytisine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monotherapy (Cytisine only) (Active Comparator): 12 weeks of cytisine: Participants allocated cytisine will be instructed to follow the manufacturer's 25-day dosing regimen, then follow a maintenance dose of cytisine from day 26 to week 12. Participants will also receive six months of text-based smoking cessation support.
  Interventions: Drug: Cytisine
- Monotherapy (Nicotine e-cigarette only) (Active Comparator): 12 weeks of a nicotine e-cigarette. Participants will also receive six months of text-based smoking cessation support.
  Interventions: Drug: Nicotine delivered via an e-cigarette
- Combination therapy (Cytisine plus a nicotine e-cigarette) (Active Comparator): 12 weeks of cytisine (as above) and 12 weeks of a nicotine e-cigarette. Participants will also receive six months of text-based smoking cessation support.
  Interventions: Combination Product: Cytisine plus nicotine delivered via an e-cigarette

INTERVENTIONS:
Drug: Cytisine — Standard dosing of:
  * days 1-3: one tablet (1.5mg) every two hours through the waking day (six tablets/day)
  * days 4-12: one tablet every 2.5 hours (five tablets/day). Quit smoking date is day five.
  * days 13-16: one tablet every three hours (four tablets/day)
  * days 17-20: one tablet every 4-5 hours (three tablets/day)
  * days 21-25: one tablet every six hours (two tablets/day)
  Followed by a maintenance dose of cystine from day 26 to week 12 (one tablet every six hours: two tablets/day)
  Other Names: Brand name: Tabex
  Arms: Monotherapy (Cytisine only)
Drug: Nicotine delivered via an e-cigarette — Pod device delivering nicotine. Nicotine strength: 30mg/ml (3%). Flavour: Tobacco
  Other Names: Brand name: UpOx
  Arms: Monotherapy (Nicotine e-cigarette only)
Combination Product: Cytisine plus nicotine delivered via an e-cigarette — Cytisine: Standard dosing of:
  * days 1-3: one tablet (1.5mg) every two hours through the waking day (six tablets/day)
  * days 4-12: one tablet every 2.5 hours (five tablets/day). Quit smoking date is day five.
  * days 13-16: one tablet every three hours (four tablets/day)
  * days 17-20: one tablet every 4-5 hours (three tablets/day)
  * days 21-25: one tablet every six hours (two tablets/day)
  Followed by a maintenance dose of cystine from day 26 to week 12 (one tablet every six hours: two tablets/day)
  Nicotine e-cigarette: Pod device delivering nicotine. Nicotine strength: 30mg/ml (3%). Flavour: Tobacco
  Other Names: Brand names: Tabex and UpOx
  Arms: Combination therapy (Cytisine plus a nicotine e-cigarette)

SUMMARY:
This research focuses on maximizing the benefits of proven smoking cessation interventions to support people who smoke to quit, as part of the strategy to help New Zealand become smoke-free. A large, pragmatic community-based clinical trial is planned which draws on 15 years of smoking cessation research undertaken by the study team. This research has shown that both cytisine and nicotine e-cigarettes are more effective than nicotine replacement therapy at helping people to quit smoking, and are more acceptable to users. New Zealand research has also shown that text-messages offering advice and support around quitting smoking are highly effective and acceptable. The planned trial will test whether using cytisine and nicotine e-cigarettes together will help more New Zealanders to quit smoking long-term, compared to using cytisine alone or nicotine e-cigarettes alone. Participants in all three groups will also receive smoking cessation text-messaging behavioral support.

DETAILED DESCRIPTION:
Aim:

To evaluate the effectiveness, safety, and acceptability of combination treatment (cytisine plus nicotine e-cigarettes) compared to monotherapy (cytisine only or nicotine e-cigarettes only) on six-month smoking abstinence.

Trial design:

A single-blind, pragmatic three-arm, parallel group, pragmatic, community-based randomized trial.

Eligibility criteria:

Eligible participants must be daily smokers who live in New Zealand, are aged ≥18 years, and have no contraindications to the study treatment. Participants must be motivated to quit smoking within the next two weeks, be able to provide online consent, have daily access to a mobile telephone that can text and have access to the internet via a computer or smart phone. Participants must also be willing to use cytisine or an e-cigarette or both products to help quit smoking. Full details of inclusion and exclusion criteria are provided later in this trial registration.

Recruitment:

Participants will be recruited from throughout New Zealand using multi-media advertising, with targeted promotion to reach indigenous Māori, Pacific and low socio-economic groups given their disproportionately higher smoking prevalence. Advertisements will direct potential participants to a trial website where they can read the participant information sheet. A two step-consent process will be used. First, interested participants will be asked for on-line consent to complete an online screening questionnaire to determine their eligibility for the trial and verify their phone number. Second, eligible and interested participants will then provide online consent to enter the trial.

Baseline information:

Baseline data will then be collected via the online platform, and will include: demographic data, smoking history, cigarette dependence, motivation to quit, withdrawal symptoms and craving, cannabis use, alcohol use, self-reported comorbidities, concomitant medication, and health-related quality of life. Full details on the baseline data are provided later in this trial registration. The participant will then be asked to click the 'randomization' button, whereupon they will be immediately randomized and informed of their allocated intervention.

Randomization:

Participants will be assigned a unique registration number allocated by a central computer, following details submitted via the study website. Eligible participants will be randomized via computer (3:3:2 ratio) to one of three trial groups using stratified block randomization (block sizes of eight), and stratified by ethnicity (Māori, non-Māori). The randomization sequence will be generated by the trial statistician, and centrally managed and concealed until the point of randomization.

Blinding:

This is a single-blind trial as participants will be aware of the intervention to which they have been allocated, and data collection by the trial research assistants will include questions specific to use of participants allocated treatment. Except for the trial statistician, the trial steering committee members will remain blinded to treatment allocation until analyses are complete. The statistical analysis plan will be finalized and uploaded to the trial registry prior to the first participant being randomised.

Interventions:

Participants will be randomized to either 12 weeks of: 1) cytisine plus nicotine e-cigarette, 2) cytisine; or 3) nicotine e-cigarette. Participants allocated cytisine will be instructed to follow the manufacturer's 25-day dosing regimen. However, a maintenance dose of cytisine will be added for day 26 to week 12. Full details of the dosing regimen are provided later in this trial registration. Participants allocated a nicotine e-cigarette will be instructed to follow the manufacturer's instructions for use, with ad libitum use over 12 weeks. The e-cigarette device used in the trial will be the 'UpOX', a closed pod system with a 3% nicotine salt (30mg/mL). A tobacco flavour e-liquid will be provided as this is the usual flavour chosen by smokers when they are transitioning away from tobacco. Participants will be advised that they should try and use only the product provided, but if they are finding the nicotine strength is not sufficiently addressing their carvings (or the flavour is distasteful) they are free to try alternative nicotine strengths or flavours, but that this will be at their own cost). Participants will be asked at follow-up about any switching of products. Participants allocated both cytisine and a nicotine e-cigarette will be instructed to follow the manufacturer's instructions for use (as mentioned above). All participants will also receive a evidence-based, text-message behavioral support program. This theoretically-based text message program will provide smoking cessation advice and motivation to support individuals to quit smoking and maintain cessation. The program includes 2-way functionality to support individuals during cravings. Regular, text messages providing smoking cessation advice, tips to cope with cravings, advice on avoiding smoking triggers, and motivational support will be delivered over a six-month period (five messages a day for six weeks, then three per week until the end of the 26th week - i.e., six-month follow-up). All 12-weeks of trial products will be couriered to participants immediately after randomization, at no cost to participants. The courier company will notify the study center immediately after the courier pack has been delivered, which will trigger the scheduling of the 'quit date' (day 0) follow-up call and the start of the text message behavioural support program.

Follow-up:

Participants will be asked to begin their treatment the day after they receive their courier pack and to reduce their smoking ad libitum over the first four days of treatment so that they are not smoking at all by the fifth day ('quit date'). Participants will be called on their quit date to verify they are quitting on that day (and to collect outcome data). If a participant states that they are not quitting on the scheduled 'quit date', they will be given one chance to reset their quit date within the next seven days, with this date becoming their new 'quit date' (which will trigger the scheduling of all subsequent follow-up calls). For participants who are unable to be contacted at quit date, their 'quit date' will be set in the system as six days after they received their courier pack (which will trigger the scheduling of all subsequent follow-up calls). Participants will be advised to continue with their allocated treatment irrespective of any lapses back to smoking. Further follow-up calls will be made at one, three and six months after their quit date to collect outcome data. Approximately two thirds of participants will also be contacted 12 months after their quit date to collect outcome data.

Outcome data:

The primary outcome is six-month carbon-monoxide verified continuous abstinence from smoking (i.e. smoking ≤ five cigarettes since quit date). Outcomes collected at three, six, and 12 months post-quit date include other cessation outcomes, treatment use, acceptability, and adverse events. Full details on the outcome data are provided later in this trial registration.

Trial power:

A sample size of 800 (N=300 in the cytisine group, N=300 in the cytisine plus nicotine e-cigarette group, and N=200 in the nicotine e-cigarette group) will provide 90% power at two-sided p=0.05 to detect an absolute difference of 13% in six-month smoking abstinence rates between the combination treatment group and the cytisine group, and 16% difference between the combination treatment group and the nicotine e-cigarette group (taking account of multiple testing). The predicted difference is based on trial evidence for six month verified continuous abstinence quit rates of 9% for nicotine e-cigarettes, 12% for cytisine, and 25% for combination cessation treatment (averaged). The sample size accounts for a 28% loss-to-follow-up at six months.

Statistical analysis:

All statistical analyses will be performed using SAS version 9.4 (SAS Institute Inc. Cary NC), and R. Data analyses will be specified a priori in a statistical analysis plan prepared by the trial statistician and posted on the trial registry prior to the first participant recruitment. No interim analyses will be undertaken. All analyses will be conducted for the following comparisons, 1) cytisine plus nicotine e-cigarettes vs cytisine and 2) cytisine plus nicotine e-cigarettes vs nicotine e-cigarettes. The main analyses will be carried out on an intention-to-treat basis, with multiple imputation analysis performed to account for missing data using the fully conditional specification logistic regression method (data will be assumed to be missing at random).

ELIGIBILITY:
Inclusion Criteria:

* Daily smokers who live in New Zealand
* Aged ≥18 years
* Motivated to quit smoking within the next two weeks
* Able to provide consent
* Have daily access to a mobile telephone that can text
* Have access to the internet via a computer or smart phone
* Are willing to use cytisine or an e-cigarette or both products to help quit smoking

Exclusion Criteria:

* Have another person in their household currently enrolled in the study
* Are pregnant/breastfeeding, or are women trying to become pregnant in the next three months
* Are currently using smoking cessation medication (including using e-cigarettes daily for the last month)
* Are enrolled in another cessation programme/trial
* Have a known hypersensitivity to cytisine or nicotine e-cigarettes
* Self-report moderate/severe renal impairment
* Are undergoing treatment for active/latent tuberculosis
* Have experienced a myocardial infarction, stroke, or severe angina within the previous two weeks
* Have uncontrolled high blood pressure (>150 mmHg systolic, >100 mmHg diastolic)
* Have a history of seizures / epilepsy
* Have a strong preference to use or not to use cytisine and/or e-cigarettes in their quit attempt.
* Have a history of severe allergy and/or poorly controlled asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with verified continuous smoking abstinence | Six months post-quit date
  Defined as self-report of smoking not more than five cigarettes from the Quit date (day 0) and confirmed by standardized exhaled carbon-monoxide (CO) measurement with a Bedfont Smokerlyzer, (≤9 ppm signifying abstinence). Sensitivity analysis will be undertaken looking at different cut-offs for the CO measurement, given lack of consensus about the best reading to use.

SECONDARY OUTCOMES:
Age | Assessed at baseline
  Date of birth will be recorded to enable the age at baseline to be reported for each treatment group (presented as a mean, with the associated standard deviation)
Gender | Assessed at baseline
  Gender will be reported as the proportion of male, female, and gender diverse at baseline, for each treatment group
Ethnicity (self-reported) | Assessed at baseline
  Ethnicity will be reported as the proportion of Maori, Pacific or Other at baseline, for each treatment group.
Education | Assessed at baseline
  Education level will be reported as the proportion of participants with "less than 12 years of schooling" or "equal or more than 12 years of schooling" or "refuse to answer" at baseline, for each treatment group.
Age started smoking | Assessed at baseline
  The age participants started smoking will be reported, with results presented as a mean (with the associated standard deviation) for each treatment group.
Number of years of continuous smoking | Assessed at baseline
  Participant's will be asked how many years they have been smoking continuously, with results presented as a mean (with the associated standard deviation) for each treatment group.
Type of cigarettes smoked | Assessed at baseline
  Type of cigarettes smoked will be reported as the proportion smoking factory-made only, roll-your-own tobacco only or both at baseline, for each treatment group
Number of cigarettes smoked per day | Assessed at baseline
  The number of cigarettes smoked per day will be asked, with results presented as a mean (with the associated standard deviation) for each treatment group.
Mean pack size (Factory-made cigarettes) | Assessed at baseline
  Participants who smoke factory-made cigarettes will be asked what pack size they normally purchase (e.g. Pack of 20) with results presented as a mean (with the associated standard deviation) for each treatment group.
Median pack size (Factory-made cigarettes) | Assessed at baseline
  Participants who smoke factory-made cigarettes will be asked what pack size they normally purchase (e.g. Pack of 20), with results presented as a median (with the associated interquartile range) for each treatment group.
Mean pouch size (Roll your-own tobacco) | Assessed at baseline
  Participants who smoke roll your-own tobacco will be asked what pouch size they normally purchase (e.g. Pack of 20) with results presented as a mean (with the associated standard deviation) for each treatment group.
Median pouch size (Roll your-own tobacco) | Assessed at baseline
  Participants who smoke roll your-own tobacco will be asked what pouch size they normally purchase (e.g. Pack of 20), with results presented as a median (with the associated interquartile range) for each treatment group.
Time taken to smoke the contents of a pack or pouch | Assessed at baseline
  Participants will be asked how many days it takes for them to smoke the contents of a pack or pouch, with results presented as a mean (with the associated standard deviation) for each treatment group.
Level of cigarette dependence | Assessed at baseline
  The level of cigarette dependence will be determined using the Heaviness of Smoking Index (HSI), which is a two-item measure based on: 1) the number of cigarettes smoked per day (cpd), categorized as: 10 or fewer cpd = 0 points; 11-20 cpd = 1 point; 21-30 cpd = 2 points; 31 cpd or more = 3 points), and 2) the time to first cigarette of the day, categorized as: within 5 minutes = 3 points, 6-30 minutes = 2 points; 31-60 minutes = 1 point; More than 60 minutes = 0 points. The HSI total score is calculated by summing these two items and has a range of 0 to 6, where higher scores indicate greater dependence. The proportion of participants with low cigarette dependence (total scores: 0-2), moderate cigarette dependence (total scores:3-4) and high cigarette dependence (total scores: 5-6) will be reported for each treatment group.
At least one quit attempt in the past 12 months | Assessed at baseline
  The proportion of participants who report at least one quit attempt in the past 12 months, will be reported for each treatment group.
Time quit, for last quit attempt | Assessed at baseline
  Of those who report at least one quit attempt in the past 12 months, the longest time participants managed to stop smoking for (in days) will be reported, with results presented as a median (with the associated interquartile range) for each treatment group.
Methods used in previous quit attempt | Assessed at baseline
  Of those who report at least one quit attempt in the past 12 months, the proportion reporting use of particular methods they used will be summarized for each treatment group. Methods will include nicotine patches, nicotine gum, nicotine lozenges, nicotine mouth spray, zyban (buproprion), nortriptyline (norpress), varenicline (champix), Quitline, community-based smoking cessation services, nicotine e-cigarette (vape), nicotine-free e-cigarette (vape), nothing, and other (free text option).
Reduction in the number of cigarettes smoked in the past 12 months | Assessed at baseline
  The proportion of participants who have cut down on the number of cigarettes they smoked in the past 12 months will be reported as "Yes" or "No" for each treatment group.
Motivation to quit | Assessed at baseline
  Motivation to quit in the next two weeks will be measured using a five point Likert Scale (where 1=not very motivated and 5=very motivated), with results presented as a mean (with the associated standard deviation) for each treatment group.
Chances of giving up smoking | Assessed at baseline
  Chances of giving up smoking for good this time, will be measured using a five point Likert Scale (where 1=extremely low and 5=extremely high), with results presented as a mean (with the associated standard deviation) for each treatment group.
Living with other people who smoke tobacco | Assessed at baseline
  The proportion of participants living with other people who smoke tobacco will be reported as "Yes", "No", or "Sometimes" for each treatment group
Living with other people who use nicotine e-cigarettes (vapes) | Assessed at baseline
  The proportion of participants living with other people who use nicotine e-cigarettes (vapes) will be reported as "Yes", "No", or "Sometimes" for each treatment group.
Has close friends who use nicotine e-cigarettes (vapes) | Assessed at baseline
  The proportion of participants living with close friends who use nicotine e-cigarettes (vapes) will be reported as "Yes" or "No" for each treatment group.
Alcohol use | Assessed at baseline
  Alcohol use will be measured using the three item Alcohol Use Disorders Identification Test (AUDIT-C). Item 1 asks "How often have you had a drink containing alcohol in the past year" with options of: Never (score=0); Monthly or less (score=1); 2-4 times per month (score=2); 2-3 times per week (score=3); 4 or more times a week (score=4). Item 2 asks "How many drinks do you usually have if you are drinking" with options of: 1 or 2 (score=0); 3 or 4 (score=1); 5 or 6 (score=2); 7 to 9 (score=3); 10 or more (score=4). Item 3 asks "How often have you had six or more drinks on one occasion in the past year?" with options of: Never (score=0); Less than monthly (score=1); Monthly (score=2); Weekly (score=3); Daily or almost daily (score=4). A total score ranges from 0 to 12. Higher scores indicate greater risk of alcohol dependence. Results will be presented as a mean (with the associated standard deviation) for male, female and gender diverse for each treatment group.
Cannabis use | Assessed at baseline
  Participants will be asked if they have used cannabis for recreational or non-medical purposes in the last 12 months, shown as the percentage reporting 'Yes' or 'No'.
Self-reported continuous smoking abstinence | Assessed at one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as the proportion of participants who self-report smoking not more than five cigarettes, reported by treatment group
Self-reported 7-day point prevalence smoking abstinence | Assessed at one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as the proportion of participants who self-report having smoked no cigarettes (not even a puff) in the past seven days, reported by treatment group
Change from baseline in the number of cigarettes smoked per day (if smoking) by participants | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Number of cigarettes smoked per day (if smoking) by participants, presented as summary statistics (mean, median, standard deviation, IQR)
Reduction in smoking by participants | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as reducing cigarette consumption by at least 25% in terms of numbers of cigarettes smoked per day
Time to first lapse back to smoking by participants | Assessed at one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as time to first cigarette smoked from the quit date, even a single puff
Time to first relapse back to smoking by participants | Assessed at one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as time to smoking more than five cigarettes a day for three or more days in a row.
Proportion of participants who use other smoking cessation methods | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked about the use of NRT and other nicotine products, and non-NRT methods of cessation such as Zyban (buproprion), clonidine, nortriptyline, varenicline, acupuncture, Quitline etc.
Health-related quality of life (five domains) | Assessed at baseline, three, six and 12 months post-quit date
  Measured using the EQ-5D-5L - a standardized measure of health-related quality of life developed by the EuroQol Group. EQ-5D-5L is not an abbreviation. The EQ-5D-5L consists of five questions - each describe a different dimension of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems. moderate problems, severe problems, extreme problems (labelled 1-5). Answers will be valued (weighted to New Zealand population norms) and transformed into a utility score using a scoring algorithm, and presented as a mean (with the associated standard deviation) for each treatment group.
Health-related quality of life (self-rated health) | Assessed at baseline, three, six and 12 months post-quit date
  The EQ-5D-5L also includes a visual analogue scale, where the respondent records their self-rated health on a 1-100 scale where the endpoints are labelled 'The best health you can imagine' (labelled 100) and 'The worst health you can imagine' (labelled 0). The EQ VAS score will be summarized using the mean (and the associated standard deviation) by treatment group.
Participant compliance with cytisine use | Measured at three months post quit date.
  Defined as having taken ≥80% of the required number of tablets over the three-month intervention period.
Number of cytisine tablets taken by participants | Measured at one and three months post quit date.
  Based on number of pills remaining, to be reported for each cytisine treatment group (presented as a mean, with the associated standard deviation)
Daily use of the allocated treatment by participants | Measured at quit date (day 0), then at one month post quit date.
  Proportion of participants who are currently using the allocated treatment (Yes/No), reported by treatment group
Reasons for not using allocated treatment | Measured at quit date (day 0), then at one month post quit date.
  Proportion of participants who report any given reason for non-use of treatment, reported according to treatment group
Frequency of use of the e-cigarette, by participants allocated e-cigarettes | Measured at three months post quit date.
  Participants allocated e-cigarettes will be asked how often they currently vape, with answer options of: not at all; daily; every couple of days; at least weekly; or other (free text option). The proportion of participants answering each option will reported according to each treatment group that received e-cigarettes.
Number of nicotine pods used, by participants allocated e-cigarettes | Measured at one and three months post quit date.
  Based on number of pods remaining to be reported for each e-cigarette treatment group (presented as a mean, with the associated standard deviation)
Signs and symptoms of nicotine withdrawal in participants | Measured at baseline and at three months (end of treatment).
  Measured using the Mood and Physical Symptoms Scale (MPSS) which consists 5-point ratings of depressed mood, irritability, restlessness, hunger and difficulty concentrating. The MPSS score is calculated by summing all 5 items (scored 1-5: not at all, slightly, moderately, very, extremely) and has a range of 5 to 25, where higher scores indicate greater nicotine withdrawal. Scores will be presented as a mean with the associated standard deviation, for each treatment group.
Urge to smoke in participants | Measured at baseline and at three months (end of treatment).
  Measured using a 6-point rating of time spent with an urge to smoke (scored 0-5: not at all, a little of the time, some of the time, a lot of the time, almost all of the time, all of the time), and the strength of these urges over the past week (scored 0-5: no urges, slight, moderate, strong, very strong, extremely strong). Participants who tick 'Not at all' for time spent with urges to smoke, then skip to the next section of questions and don't answer the question on strength of urges. For these participants the strength of urges is set at 0, therefore, this question will then have values 0 to 5. The urge score is calculated by summing the two urges questions and has a range 0 to 10, where higher scores indicate greater urge to smoke. Scores will be presented as a mean with the associated standard deviation, for each treatment group.
Treatment switching (crossover from cytisine-only to e-cigarette) | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants allocated cytisine only, will be asked if they accessed and used an e-cigarette during the trial, with results reported as the proportion at each time period.
Treatment switching (crossover from cytisine-only to e-cigarette): nicotine content of e-cigarette | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants allocated cytisine only, who accessed and used an e-cigarette during the trial will be asked if the device had nicotine in it or not, with results reported as proportions at each time period
Treatment switching (crossover from e-cigarette-only to cytisine) | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants allocated e-cigarettes only will be asked whether they accessed and used cytisine during the trial, with results reported as proportions at each time period.
Treatment switching (crossover from e-cigarette-only to cytisine): source of cytisine | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants allocated e-cigarettes-only, who accessed (but were not allocated) cytisine, will be asked how they obtained the cytisine, with results reported as proportions for each stated option at each time period.
Change in e-cigarette use | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants allocated to the e-cigarette groups will be asked whether they changed the type of e-cigarette device and/or the nicotine strength and/or flavour they used in the e-cigarettes provided. If they did, they will be asked when they did this, and what the device type, nicotine strength and/or flavour was.
Dual use of treatment and tobacco by participants | Assessed at one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Defined as daily use of both the allocated treatment and continued daily smoking of cigarettes.
Continuation of product use by participants | Measured at six (in all) and 12 months (in a subsample).
  Defined as continued use of the allocated treatment by participants after the end of the designed three-month treatment period.
Acceptability of allocated product | Measured at three months post-quit date (end of treatment)
  Participants will be asked for their views on the use of the allocated product as a cessation aid, that is what participants liked or disliked about using the product(s): Answers will be provided as free text.
Participants recommendations regarding the allocated product | Measured at three months post-quit date (end of treatment)
  Participants will be asked if they would recommend the allocated treatment to another person who smoked but wanted to quit.(answer options of: Yes; No; Did not use product).
Number of participants with self-reported adverse events | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked about any new, unusual, unexpected health events during or since starting treatment, and whether they felt they were related to treatment. Serious adverse events will be classified as non-serious or serious (death, life threatening, hospitalization, persistent or sustained disability/incapacity, congenital abnormality/birth defect, significant medical event). The likelihood of causality will be assessed using the World Health Organization Standardized Case Causality Assessment Tool (certain, probable/likely, possible, unlikely, conditional/unclassified, unassessable/unclassifiable).
Number of self-reported adverse events | Assessed at quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked about any new, unusual, unexpected health events during or since starting treatment, and whether they felt they were related to treatment. Serious adverse events will be classified as non-serious or serious (death, life threatening, hospitalization, persistent or sustained disability/incapacity, congenital abnormality/birth defect, significant medical event). The likelihood of causality will be assessed using the World Health Organization Standardized Case Causality Assessment Tool (certain, probable/likely, possible, unlikely, conditional/unclassified, unassessable/unclassifiable).
Change from baseline in body mass index | Asked at three and six months post-quit date
  Self-reported height (in cm) and weight (kg) will be measured at baseline and combined to determine baseline body mass index (kg/m2). Self-reported weight (kg) will be asked at three and six months to determine change in body mass index from baseline to three and six months in those participants that have quit smoking at these timepoints, compared to those that have not quit smoking.
Change from baseline in frequency of shortness of breath in participants | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Self-reported frequency of shortness of breath will be measured at baseline (How often do you get short of breath? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Self-reported frequency of shortness of breath will be re-assessed at follow-up using the same criteria to determine change in frequency of shortness of breath from baseline to three and six months post quit (and at 12 months post-quit date in a subsample).
Change from baseline in frequency of coughing in participants | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Self-reported frequency of coughing will be measured at baseline (How often do you cough? Response options are: Not at all; A little of the time; Some of the time; A lot of the time; All of the time). Self-reported frequency of coughing will be re-assessed at follow-up using the same criteria, to determine change in frequency of coughing from baseline to three and six months post quit (and at 12 months post-quit date in a subsample).
Change from baseline in asthma severity, in those participants with asthma | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked at baseline if have have asthma (self-reported: Yes/No). Participants who report that they do have asthma will be asked at follow-up whether their asthma has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study.
Change from baseline in severity of chronic pain, in those participants with chronic pain. | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked at baseline if have have chronic pain (self-reported: Yes/No). Participants who report that they do have chronic pain will be asked at follow-up whether their chronic pain has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study.
Change from baseline in severity of Chronic Obstructive Pulmonary Disease (COPD), in those participants with COPD. | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked at baseline if have have COPD (self-reported: Yes/No). Participants who report that they do have COPD will be asked at follow-up whether their COPD has been: much worse; a bit worse; about the same; a bit better; or much better since starting the study.
Change from baseline in severity of mental health concerns, in those participants with mental health concerns. | Measured at three and six months post-quit date (and at 12 months post-quit date in a subsample)
  Participants will be asked at baseline if they are currently receiving treatment for any mental health concerns (self-reported: depression; schizophrenia or related disorder; anxiety; another mental health concern ). Participants who report that they are currently receiving treatment for any mental health concerns will be asked at follow-up whether their mental health symptoms have been: much worse; a bit worse; about the same; a bit better; or much better since starting the study.
Concomitant medication | Assessed at baseline, quit date (day 0), then one, three, and six months post-quit date (and at 12 months post-quit date in a subsample)
  Information about types of medication currently used
Mean number of text-based behavioral support messages received by participants | Assessed at six months
  Number of text-based behavioral support messages received by participants during the six months, reported as a mean, with associated standard deviation
Median number of text-based behavioral support messages received by participants | Assessed at six months
  Number of text-based behavioral support messages received by participants during the six months, reported as a median, with associated interquartile range
Marginal cost per quitter | Assessed at six months
  If combination treatment is better than monotherapy, a cost-effectiveness analysis will be undertaken. The total number of cigarettes smoked between quit date (QD) and 6-month follow-up (FU) will be multiplied by the mean cigarette cost. The total number of cytisine tablets used by participants between QD and 6-month FU will be multiplied by the tablet cost. The total number of e-cigarette pods used by participants between QD and 6-month FU will be multiplied by the pod cost. The total cost will be the sum of the above. The cost-per-quitter will be the total cost by quit status (using self-reported continuous smoking abstinence). The incremental cost-effectiveness ratio will be the total cost and quitting status. The cost-per-person reducing their daily cigarette consumption will be assessed by crossing the total cost by a binary variable created for the reduction of at least 25% in the number of cigarettes smoked per day between QD and 6-month FU.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- National Institute for Health Innovation, School of Population Health, Faculty of Medical and Health Sciences, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
This plan is currently being developed and will be made available soon.
  Please note that at least 25% of trial participants are likely to be Indigenous Māori. In New Zealand "indigenous data sovereignty recognizes that Māori data should be subject to Māori governance. Māori data sovereignty supports tribal sovereignty and the realization of Māori and Iwi aspirations." Requests to access trial data provided by Māori participants will be reviewed and considered by the Māori Research Advisory Committee at the National Institute for Health Innovation, University of Auckland.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting nine months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Requests for access to individual participant data, or trial documents, will be considered where: 1) the request is from qualified researchers engaging in independent scientific research; 2) the proposed use aligns with public good purposes; 3) a research proposal and Statistical Analysis Plan are provided for review and approval; 4) the request does not conflict with other requests or planned use by members of the trial steering committee; and 5) the requestor is willing to sign a data access agreement. Please send all requests to the principal investigator.

REFERENCES:
- [Derived] Walker N, Calder A, Barnes J, Laking G, Parag V, Bullen C. Effectiveness of nicotine salt vapes, cytisine, and a combination of these products, for smoking cessation in New Zealand: protocol for a three-arm, pragmatic, community-based randomised controlled trial. BMC Public Health. 2023 Sep 11;23(1):1760. doi: 10.1186/s12889-023-16665-w. PMID 37697327

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT05311085/SAP_000.pdf